CLINICAL TRIAL: NCT03241095
Title: The Efficacy of Osteopathic Manipulative Treatment (OMT) on the Swing Via Objective Data From Golf Simulator Swing Analysis and Subjective Data
Brief Title: The Efficacy of Osteopathic Manipulative Treatment (OMT) on the Golf Swing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMCH-2017-25925
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Manipulation, Osteopathic
Keywords: Osteopathic Manipulation Treatment; Golf
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Sham OMT (Sham Comparator)
  Interventions: Procedure: Sham intervention
- OMT (Active Comparator)
  Interventions: Procedure: OMT (Osteopathic Manipulative Treatment)

INTERVENTIONS:
Procedure: OMT (Osteopathic Manipulative Treatment) — The co-hort will receive OMT. Each participant will perform 10 swings golf swings to determine a baseline measure the strength of their golf swing. This co-hort will then be evaluated by the physician and be given OMT.
  Arms: OMT
Procedure: Sham intervention — The co-hort participants will each perform 10 swings golf swings to determine a baseline measure the strength of their golf swing. Theythen be given a sham OMT procedure.
  Arms: Sham OMT

SUMMARY:
The purpose of the study is to investigate if osteopathic manipulative treatment (OTM) improves the golf swing of the participants. Study participants will be randomized into three groups, we will stratify by age and gender to make them as uniform as possible. One group will receive no intervention other than a 10-minute break between the pre and post measurements. A second group will receive a sham intervention where the doctor will pretend to give the participant OTM. The third group will receive real OTM.

Participants will perform a sample of 10 golf swings pre and post intervention which will be measured by a golf simulator. They will also complete a brief health history and pre/post self-evaluation of their swing.

ELIGIBILITY:
Inclusion Criteria: Adult golfers (18 years old or over) -

Exclusion Criteria: Anyone under 18 years, people that do not golf.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Strength of golf swing as measured by the carry distance (the distance the ball flies in the air) | 30 minutes
  The participant will perform 10 swings into a golf simulator using a 5 iron. The simulator will record the information for each swing. Measurements include: Club head speed (Mph), Ball speed (Mph), Launch angle (Deg), Azimuth (Deg), Side spin (Rpm), Back spin (Rpm), Total spin (Rpm), Descent angle (Deg), Carry (Yds),Total distance (Yds), Offline (Yds), Peak height (Yds). We will be looking at the 'Carry' variable, before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Buffington, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Mayo Clinic Health System - Family Medicine Clinic, Mankato, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No